CLINICAL TRIAL: NCT04938648
Title: Align: Aligning Medications With What Matters Most
Brief Title: Aligning Medications With What Matters Most
Acronym: ALIGN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Kaiser Permanente (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00286353; 5U54AG063546-02 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-24 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Polypharmacy; Alzheimer Disease and Related Dementias
Keywords: Deprescribing
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Patient and care partner dyads are randomly assigned to receive the pharmacist-led intervention immediately after an educational mailing or to a delayed intervention control group that will receive the pharmacist-led component 3 months after the mailing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of the following:
  1. mailing deprescribing educational materials to care partners and people living with dementia (PLWD);
  2. dyads will receive a telehealth visit with a clinical pharmacist to discuss the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences;
  3. pharmacist- primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations to the PCP.
  Interventions: Behavioral: Pharmacist-led deprescribing intervention
- Delayed Intervention (wait list control) (Active Comparator): The delayed intervention consists of the following:
  1. mailing deprescribing educational materials to care partners and people living with dementia (PLWD);
  2. three months after mailing the deprescribing educational materials, dyads will receive a telehealth visit with a clinical pharmacist to discuss the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences.
  3. pharmacist- primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations to the PCP.
  Interventions: Behavioral: Pharmacist-led deprescribing intervention

INTERVENTIONS:
Behavioral: Pharmacist-led deprescribing intervention — 1) direct-to-consumer deprescribing educational materials designed to activate the care partner and people living with dementia PLWD; 2) a telehealth visit in which a clinical pharmacist discusses benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences; and 3) pharmacist-PCP communication in which the pharmacist provides tailored deprescribing recommendations designed to be useful and actionable for the PCP

SUMMARY:
The Aligning Medications with What Matters Most (ALIGN) study will assess the feasibility and preliminary efficacy of a deprescribing intervention to reduce medication regimen complexity and treatment burden for people living with dementia (PLWD) and their care partners.

DETAILED DESCRIPTION:
People living with dementia (PLWD) use more medications and have more complex medication regimens than people without dementia. Medication regimen complexity is a major source of burden for family caregivers of PLWD and has been associated with numerous adverse outcomes. Therefore, the investigators propose a novel intervention, ALIGN: Aligning Medications with What Matters Most, to optimize prescribing and reduce medication regimen complexity by focusing on what matters most to the patient and caregiver, beyond rigid adherence to clinical practice guidelines. ALIGN is informed by learnings from OPTIMIZE, the investigator team's patient-centered, pragmatic deprescribing intervention for PLWD in primary care that is currently being prospectively evaluated. OPTIMIZE consists of a patient-level intervention comprised of a deprescribing educational brochure, and a clinician-level intervention comprised of a deprescribing educational session for primary care providers (PCPs), deprescribing "tip sheets" and clinic-level feedback on rates of potentially inappropriate medication prescribing in PLWD. ALIGN builds on OPTIMIZE by more explicitly addressing the informational and decisional needs of caregivers through a shared decision making process facilitated by clinical pharmacists. The investigators propose a pilot study to assess the feasibility and acceptability of ALIGN in two different health care systems, and to identify the most appropriate primary outcome measure for a subsequent embedded pragmatic trial (ePCT). Target enrollment is 60 patient-care partner dyads. Patients will be aged ≥65 years with dementia and >5 chronic medications. Primary outcomes are intervention feasibility and acceptability among patients, care partners and PCPs; and feasibility of the patient-level Medication Regimen Complexity Index and Family Caregiver Medication Administration Hassles Scale at baseline and 3 months. Findings from this pilot study will guide the design, implementation and subsequent evaluation of ALIGN in an ePCT, laying the groundwork to reduce medication regimen complexity and burden for PLWD and their caregivers in diverse primary care settings.

This proposed pragmatic intervention has the following aims:

Specific Aim 1: To assess the feasibility and acceptability of ALIGN in two different health care systems, to guide the subsequent evaluation of the effectiveness of the intervention in an embedded pragmatic trial (ePCT).

Specific Aim 2: To determine the feasibility of the primary and secondary outcome measures for the subsequent ePCT.

1. To determine the feasibility of measuring the primary outcome, the patient-level Medication Regimen Complexity Index (pMRCI), within the existing electronic health record (EHR) systems, and to compare it with a more pragmatic measure, chronic medication count, as the primary outcome measure for the ePCT.
2. To determine the feasibility of measuring the secondary outcome, the Family Caregiver Medication Administration Hassles Scale (FCMAHS), a caregiver-reported outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or greater
* Diagnosis of dementia from International Classification of Diseases (ICD) -9 or ICD-10 codes
* At least one other chronic condition
* Five or more chronic medications (to include all prescription and over-the-counter medications, both scheduled and as needed)
* Have a primary care physician at the pilot clinic who has enrolled in the study; this will be defined as having had at least 1 previous visit with that physician

Care partners:

- Family or other companions age 21 years or greater who regularly help the patient with managing medications

Exclusion Criteria:

* As both the pilot and the planned pragmatic trial will be based in primary care, individuals residing in long term care facilities or enrolled in hospice will be excluded.
* Individuals who cannot converse comfortably in English will be excluded because the FCMAHS has not been validated in other languages.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Green, MD, MPH, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Kaiser Permanente, Aurora, Colorado
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

REFERENCES:
- [Background] Boyd CM, Darer J, Boult C, Fried LP, Boult L, Wu AW. Clinical practice guidelines and quality of care for older patients with multiple comorbid diseases: implications for pay for performance. JAMA. 2005 Aug 10;294(6):716-24. doi: 10.1001/jama.294.6.716. PMID 16091574
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Background] Lin PJ, Fillit HM, Cohen JT, Neumann PJ. Potentially avoidable hospitalizations among Medicare beneficiaries with Alzheimer's disease and related disorders. Alzheimers Dement. 2013 Jan;9(1):30-8. doi: 10.1016/j.jalz.2012.11.002. PMID 23305822
- [Background] Kelley AS, McGarry K, Gorges R, Skinner JS. The burden of health care costs for patients with dementia in the last 5 years of life. Ann Intern Med. 2015 Nov 17;163(10):729-36. doi: 10.7326/M15-0381. Epub 2015 Oct 27. PMID 26502320
- [Background] Willson MN, Greer CL, Weeks DL. Medication regimen complexity and hospital readmission for an adverse drug event. Ann Pharmacother. 2014 Jan;48(1):26-32. doi: 10.1177/1060028013510898. Epub 2013 Nov 5. PMID 24259639
- [Background] Bayliss EA, Shetterly SM, Drace ML, Norton J, Green AR, Reeve E, Weffald LA, Wright L, Maciejewski ML, Sheehan OC, Wolff JL, Gleason KS, Kraus C, Maiyani M, Du Vall M, Boyd CM. The OPTIMIZE patient- and family-centered, primary care-based deprescribing intervention for older adults with dementia or mild cognitive impairment and multiple chronic conditions: study protocol for a pragmatic cluster randomized controlled trial. Trials. 2020 Jun 18;21(1):542. doi: 10.1186/s13063-020-04482-0. PMID 32552857
- [Background] Group Health Research Institute. The Chronic Care Model. Available at http://www.improvingchroniccare.org/index.php?p=CCM_Gallery&s=149. Accessed August 21, 2020
- [Background] George J, Phun YT, Bailey MJ, Kong DC, Stewart K. Development and validation of the medication regimen complexity index. Ann Pharmacother. 2004 Sep;38(9):1369-76. doi: 10.1345/aph.1D479. Epub 2004 Jul 20. PMID 15266038
- [Background] Travis SS, Bernard MA, McAuley WJ, Thornton M, Kole T. Development of the family caregiver medication administration hassles scale. Gerontologist. 2003 Jun;43(3):360-8. doi: 10.1093/geront/43.3.360. PMID 12810899

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients and care partners were enrolled as dyads. A total of 69 dyads were enrolled with available data obtained from the EHR only for the patients.
Groups:
- Intervention: The intervention consists of the following:
  1. mailing deprescribing educational materials to care partners and people living with dementia (PLWD);
  2. dyads will receive a telehealth visit with a clinical pharmacist to discuss the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences;
  3. pharmacist- primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations to the PCP.
  Pharmacist-led deprescribing intervention: 1) direct-to-consumer deprescribing educational materials designed to activate the care partner and people living with dementia PLWD; 2) a telehealth visit in which a clinical pharmacist discusses benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences; and 3) pharmacist-PCP communication in which the pharmacist provides tailored deprescribing recommendations designed to be useful and actionable for the PCP
- Delayed Intervention (Wait List Control): The delayed intervention consists of the following:
  1. mailing deprescribing educational materials to care partners and people living with dementia (PLWD);
  2. three months after mailing the deprescribing educational materials, dyads will receive a telehealth visit with a clinical pharmacist to discuss the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences.
  3. pharmacist- primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations to the PCP.
  Pharmacist-led deprescribing intervention: 1) direct-to-consumer deprescribing educational materials designed to activate the care partner and people living with dementia PLWD; 2) a telehealth visit in which a clinical pharmacist discusses benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences; and 3) pharmacist-PCP communication in which the pharmacist provides tailored deprescribing recommendations designed to be useful and actionable for the PCP
Period: Overall Study
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Started | 34 | 35
Completed | 27 | 28
Not Completed | 7 | 7
Not completed — Patient admitted to SNF hospice/LTC | 2 | 1
Not completed — Patient too ill | 0 | 1
Not completed — Patient in rehab at the time of intervention | 1 | 0
Not completed — Patient did not have memory problems | 1 | 1
Not completed — Intervention could not be scheduled within protocol window | 1 | 0
Not completed — Care partner could not be reached | 0 | 1
Not completed — Patient no longer receiving care at an eligible clinic | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were collected for patients only. Baseline data were not collected from care partners.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Delayed Intervention (Wait List Control) | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.6 (7.0) | 82.1 (8.7) | 81.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 14 | 27
  White | 14 | 18 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 10
Total number of medicines [Mean (Standard Deviation); unit: medications] | 13.1 (4.6) | 12.5 (5.5) | 12.8 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Proportion of Dyads That Opt Out of the Intervention
Description: Dyads are comprised of the person living with dementia and their care partner. We will measure the proportion of dyads that opt out of the intervention versus the dyads that agree to participate.
Time Frame: A duration of approximately 8 months
Population: This outcome is based on pre-randomization activities. The overall number of individual participants analyzed represents all potentially eligible patients identified that were further reviewed to confirm eligibility and interest in participating in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Proportion of Dyads That Opt Out of the Intervention: The intervention consists of the following:
  1. mailing deprescribing educational materials to care partners and people living with dementia (PLWD);
  2. dyads will be randomly assigned to receive a telehealth visit with a clinical pharmacist immediately after receiving the brochure or at 3 months to discuss the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences;
  3. pharmacist- primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations to the PCP.
Arm/Group | Proportion of Dyads That Opt Out of the Intervention
Number analyzed (Participants) | 424
Participants
  Excluded | 101
  Unable to reach | 122
  Declined to participate | 132
  Agreed to participate | 69

2. Primary Outcome: Feasibility as Assessed by the Number of Pharmacist Messages to the Primary Care Provider (PCP) That Receive an Acknowledgment or Response
Description: We will measure the number of pharmacist's messages that receive an acknowledgment or response from the PCP based on Electronic Medical Record (EMR) review
Time Frame: 3 months after enrollment
Population: The overall number of participants analyzed represents the number of individual participants (patients). The sample size for the treated was 34, of these 27 received the intervention, and the sample size for the control subjects was 35 of these, 28 received the intervention with available data only for those who completed the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants
  1 | 22 | 23
  2 | 4 | 4
  3 | 1 | 1

3. Primary Outcome: Feasibility as Assessed by the Number of Contacts Between Pharmacist and PCP
Description: We will measure the number of contacts between pharmacist and PCP based on Electronic Medical Record (EMR) review
Time Frame: 3 months after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants
  1 | 0 | 0
  2 | 19 | 21
  3 | 6 | 2
  ≥4 | 2 | 5

4. Primary Outcome: Feasibility as Assessed by the Number of Contacts Between Pharmacist and Dyad
Description: We will measure the number of contacts between pharmacist and PCP and dyad based on Electronic Medical Record (EMR) review
Time Frame: 3 months after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants
  1 | 0 | 1
  2 | 6 | 14
  3 | 8 | 10
  4 | 3 | 3
  ≥5 | 10 | 0

5. Primary Outcome: Feasibility as Assessed by the Direct Time Required by the Pharmacist to Complete the Intervention
Description: We will measure the amount of direct time that it takes the pharmacist to complete the intervention. We will access from pharmacist's documentation in the Electronic Medical Record (EMR).
Time Frame: 3 months after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants
  11-20 mins | 1 | 3
  21-30 mins | 7 | 11
  31-40 mins | 7 | 5
  41-50 mins | 8 | 5
  51-60 mins | 3 | 3
  61-70 mins | 1 | 0
  71-80 mins | 0 | 1

6. Primary Outcome: Feasibility as Assessed by the Indirect Time Required by the Pharmacist to Complete the Intervention
Description: We will measure the amount of indirect time that it takes the pharmacist to complete the intervention. We will access from pharmacist's documentation in the Electronic Medical Record (EMR).
Time Frame: 3 months after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants
  5-10 mins | 9 | 6
  11-20 mins | 8 | 16
  21-30 mins | 5 | 4
  31-40 mins | 0 | 2
  41-50 mins | 3 | 0
  51-60 mins | 2 | 0

7. Primary Outcome: Feasibility as Assessed by Percentage of Dyads Who Complete 2 of 2 Pharmacist Phone Calls Based on Documented Status Reports
Description: Dyads are comprised of the person living with dementia and their care partner. We will measure the percentage of dyads who complete 2 of 2 pharmacist phone calls based on documented status reports
Time Frame: Baseline and 3 months after enrollment
Population: The sample size for the treated was 34, of these 27 received the intervention, and the sample size for the control subjects was 35 of these, 28 received the intervention with available data only for those who completed the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants | 24 | 26

8. Primary Outcome: Acceptability Will be Assessed by the Acceptance Rates for the Pharmacist's Recommendations
Description: We will measure the acceptance rates for the pharmacist's recommendations as documented in the Electronic Medical Record (EMR)
Time Frame: 3 months after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 27 | 28
Participants | 23 | 24

9. Secondary Outcome: Total Medication Count
Description: We will measure the total medication count using data obtained from the EHR.
Time Frame: Baseline and 3 months after enrollment
Population: The sample size for 3-month and change measures were 27 for the treated and 28 for the control subjects with available data at 3 months.
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 34 | 35
medications
  Baseline | 13.1 (4.6) | 12.5 (5.5)
  3-month: number analyzed (Participants) | 27 | 28
  3-month | 12.6 (4.4) | 12.4 (5.4)
  Change: number analyzed (Participants) | 27 | 28
  Change | -0.6 (3.4) | -0.2 (1.7)

10. Secondary Outcome: Percentage of Participants With Data Elements Available to Calculate the Medication Regimen Complexity Index (pMRCI)
Description: The feasibility of measuring this outcome will be determined as follows: Percentage of participants with data elements available vs. unavailable to calculate the pMRCI, within the existing electronic medical record systems.
  This study assessed the feasibility of measuring the pMRCI and not actually determining the pMRCI.
  The pMRCI is a validated, widely-used tool that measures medication regimen complexity to identify patients with expected difficulty managing their regimens. Scores are derived from weighted values of regimen components (eg, dosage formulations, frequencies, and specific instructions for use). Higher scores indicate greater medication regimen complexity.
Time Frame: Baseline and 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 34 | 35
Participants
  Baseline | 34 | 35
  3-month | 27 | 28

11. Secondary Outcome: Medication Regimen Complexity Index (MRCI)
Description: The MRCI is a validated, widely-used tool that measures medication regimen complexity to identify patients with expected difficulty managing their regimens. The MRCI score is derived from weighted values of regimen components (eg, dosage formulations, frequencies, and specific instructions for use). The score has no upper limit, but higher scores indicate greater medication regimen complexity. Regimen components were combined to compute a total score and averaged.
Time Frame: Baseline and 3 months Baseline and 3 months after enrollment
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 34 | 35
score on a scale
  Baseline | 32.8 (17.5) | 29.7 (15.8)
  3-month: number analyzed (Participants) | 27 | 28
  3-month | 31.7 (22.5) | 31.7 (20.7)
  Change: number analyzed (Participants) | 27 | 28
  Change | -1.0 (12.4) | 1.2 (12.9)

12. Secondary Outcome: Response Rate for the Family Caregiver Medication Administration Hassles Scale (FCMAHS)
Description: We will measure the response rate from care partners to complete the FCMAHS over the phone or electronically.
  The FCMAHS is a validated caregiver-reported outcome measure that assesses burden associated with medication administration. The instrument consists of 24 items and four subscales: Information Seeking/Information Sharing (9 items), Safety Issues (5 items), Scheduling Logistics (7 items) and Polypharmacy (3 items). The total score range is 0-120 with higher scores indicating greater perceived hassle associated with managing some or all aspects of another person's medication regimen.
Time Frame: Baseline and 3 months after enrollment
Population: The FCMAHS was offered as an optional survey at baseline and 3 months with available data only for those who agreed to complete it. A total of 34 participants in the intervention group and 35 participants in the delayed control group were eligible to complete the survey. The sample size for the FCMAHS at baseline and 3 months are 25, 18 for the intervention group and 21, 15 for the delayed control group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 34 | 35
Participants
  Baseline | 25 | 22
  3-month | 18 | 15

13. Secondary Outcome: Time to Complete the Family Caregiver Medication Administration Hassles Scale (FCMAHS)
Description: We will measure the time it takes the care partner to complete the FCMAHS over the phone or electronically.
  The FCMAHS is a validated caregiver-reported outcome measure that assesses burden associated with medication administration. The instrument consists of 24 items and four subscales: Information Seeking/Information Sharing (9 items), Safety Issues (5 items), Scheduling Logistics (7 items) and Polypharmacy (3 items). The total score range is 0-120 with higher scores indicating greater perceived hassle associated with managing some or all aspects of another person's medication regimen.
Time Frame: Baseline and 3 months after enrollment
Population: This was an optional survey given to participants at baseline and 3 months with available data only for those who agreed to complete it. The completion rate sample size for the delayed control group at baseline was 22; data from 1 participant is missing for this variable. The sample size for the 3-month measure was 18 for the treated and 15 for the control subjects with available data at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 25 | 21
Participants
  Baseline: 0-5 mins | 11 | 8
  Baseline: 6-10 mins | 9 | 7
  Baseline: 11 or more mins | 5 | 6
  3-month: number analyzed (Participants) | 18 | 15
  3-month: 0-5 mins | 5 | 7
  3-month: 6-10 mins | 9 | 5
  3-month: 11 or more mins | 4 | 3

14. Secondary Outcome: Family Caregiver Medication Administration Hassles Scale (FCMAHS)
Description: The FCMAHS is a validated caregiver-reported outcome measure that assesses burden associated with medication administration. The instrument consists of 24 items and four subscales: Information Seeking/Information Sharing (9 items), Safety Issues (5 items), Scheduling Logistics (7 items) and Polypharmacy (3 items). The total score range is 0-120 with higher scores indicating greater perceived hassle associated with managing some or all aspects of another person's medication regimen.
Time Frame: Baseline and 3 months after enrollment
Population: This was an optional survey given to participants at baseline and 3 months with available data only for those who agreed to complete it. The completion rate sample size for the delayed control group at baseline was 22; data from 1 participant is missing for this variable. The sample size for 3 months and change measures was 18 for the treated and 15 for the control subjects with available data at 3 months.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
Number analyzed (Participants) | 25 | 21
Score on a scale
  Baseline | 33.2 (19.2) | 37.3 (25.8)
  3-Month: number analyzed (Participants) | 18 | 15
  3-Month | 29.9 (16.2) | 31.3 (23.6)
  Change: number analyzed (Participants) | 18 | 15
  Change | -3.3 (18.8) | -2.5 (14.4)

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Intervention | Delayed Intervention (Wait List Control)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 6/34 | 2/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=34) | Delayed Intervention (Wait List Control) (N=35)
Hospitalization (General disorders) | 4 | 0
ED Visit (General disorders) | 3 | 2
Observation (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04938648/Prot_SAP_000.pdf